CLINICAL TRIAL: NCT02183727
Title: L-C Ligament Versus Hamstring Autograft for Primary ACL Reconstruction: A Prospective, Randomized Controlled Trial
Brief Title: L-C Ligament Versus Hamstring Autograft for Primary ACL Reconstruction
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Data from LC1033 study of same product indicated lower than expected clinical outcomes; company, STR did not have funds to continue study.
Sponsor: Soft Tissue Regeneration, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LC1060
Record Dates: First submitted 2014-06-26; First posted 2014-07-08 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Acute Ruptures of the Anterior Cruciate Ligament
Keywords: ACL; knee injury; anterior cruciate ligament
MeSH Terms: conditions — Knee Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-C Ligament (Experimental): Soft Tissue Regeneration's L-C Ligament is an investigation, interventional device intended for ACL reconstruction surgery within 18 weeks of acute rupture of the ACL and no previous surgical treatment. The L-C Ligament temporarily replaces the human anterior cruciate ligament (ACL) and provides a bioresorbable scaffold within and around which the native ACL will regenerate over time.
  Interventions: Device: L-C Ligament
- Hamstring Autograft (Active Comparator): Hamstring autograft is the active comparator for this study. Autograft tissue is the gold-standard treatment for primary ACL reconstruction.
  Interventions: Procedure: Hamstring Autograft

INTERVENTIONS:
Device: L-C Ligament — The L-C Ligament is a bioresorbable, three-dimensional (3-D) braided scaffold made from poly L-lactic acid (PLLA) fiber. One device is used to replace the ACL. The L-C Ligament is an interventional device. The L-C Ligament is comprised of three regions: (1) The femoral tunnel attachment site, (2) The ligament region (intra-articular zone), and (3) The tibial tunnel attachment site. For several months after surgery, the L-C Ligament replaces the function of the ACL. During this time, ligament tissue regenerates within and around the L-C Ligament, which is slowly absorbed and replaced by the ACL.
  Arms: L-C Ligament
Procedure: Hamstring Autograft — The gold-standard treatment for ACL reconstruction is autograft tissue. Autograft is a piece of tendon harvested from another part of the patient's body, such as the hamstring or kneecap. In this study, the hamstring tendon from the back of the thigh of the injured (target) leg will be harvested and surgically transferred to replace the torn ACL. The attachment of the autologous tendon in the femoral and tibial bone tunnels will utilize techniques that are similar to those for the L-C Ligament. Over time the replacement tendon resorbs and a new ACL is regenerated.
  Arms: Hamstring Autograft

SUMMARY:
The purpose of this study is to compare safety and efficacy outcomes of the L-C Ligament versus Hamstring Autograft for treatment of acute rupture of the ACL.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute ruptures of the ACL who are willing to undergo treatment within 18 weeks of injury

Exclusion Criteria:

* Prior ACL reconstruction or other surgical procedure on the affected (target) knee
* Chronic ACL injury; interventional surgery scheduled 127 days or more after ACL injury
* Professional athletes currently engaged in active sport
* Prior distal femoral and/or proximal tibial fracture(s) of the target leg
* Previous or current ACL injury on contra-lateral leg
* Multi-ligament reconstruction
* Malalignment or varus thrust
* Patient > 193 cm tall (6' 4")
* The patient does not follow pre-operative rehabilitation that may have been prescribed post-injury (prior to Index Procedure)
* Confirmed connective tissue disorder
* Signs of moderate to severe degenerative joint disease
* Severe pain, swelling, or redness within 24 hours prior to surgery
* Complete or partial Posterior Cruciate Ligament (PCL) tear
* If concomitant meniscal injury is present, any of the following: 1/3rd meniscal resection; complex double-bucket tear; partially repaired meniscal tears
* Any type of lateral and/or medial meniscal tear which is not repairable (<2mm from rim)
* Additional concomitant injuries to the knee or lower extremities requiring treatment, per surgeon's discretion, that are not allowable under the Inclusion criteria
* The patient is unwilling to not participate in sporting activities for at least 9 months post-procedure
* The patient is mentally compromised
* The patient has a neuromuscular disorder that would engender unacceptable risk of knee instability, prosthesis fixation failure, or complications in postoperative care
* The patient has an active or latent infection in or about the affected knee joint or an infection site distant from the knee that may spread to the knee hematogenously
* Pregnant based on a positive beta hCG serum or an in vitro diagnostic test result or breast-feeding
* The patient is obese with a BMI > 35
* The patient has a known allergy to PLLA
* The patient has a medical condition or comorbidity that would interfere with study participation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Graft Failure | 12 Months
  Revision surgery rate at one year
Physical Knee Function measured by the IKDC | 12 Months
  Physical Knee Function at 12 Months post procedure

SECONDARY OUTCOMES:
Pain Score | Day 1
  Pain levels day 1 post-procedure
Adverse event rates | 12 months
  Rate of AEs throughout the first year of follow-up

OTHER OUTCOMES:
Physical Knee Function as measured by the Lysholm scale | over 24 months
  Physical Knee Function scores at all follow-up timepoints through Month 24
Return to Pre-Injury Physical Activity Levels as measured by the Tegner scale | over 24 months
  Physical activity level scores at all follow-up timepoints through Month 24
Knee Outcomes (Pain, symptoms, ability ot perform daily activities, sports, and quality of life) as measured by the KOOS | over 24 months
  KOOS scores at all follow-up timepoints through Month 24

CONTACTS AND LOCATIONS:
Overall Officials: Kees van Egmond, MD, Principal Investigator — Isala Klinieken, Zwolle, The Netherlands
Locations (1):
- Isala Klinieken, Zwolle, Netherlands